CLINICAL TRIAL: NCT06809192
Title: Factorial Optimization Randomized Controlled Trial to Test The Effects of Cognitive Behavioral Therapy Components For Multiple Sclerosis Fatigue
Brief Title: Factorial Optimization Trial to Test Cognitive Behavioral Therapy Components for Multiple Sclerosis Fatigue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lindsey Knowles, Assistant Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021168; K23HD111628 (NIH)
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Multiphase Optimization Strategy; Cognitive Behavioral Therapy; Relaxation; Behavioral Activation; Cognitive Therapy; Optimization; Factorial Trial
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- No Treatment (No Intervention): Participants in the "No Treatment" condition will not complete any component sessions and will complete assessments at baseline (within 1 month of randomization), at approximately 2 months after randomization (the weighted average of weeks of treatment in the other conditions), and 3-month follow-up (dated from randomization). Upon study completion, these participants will be offered the opportunity to complete a component of their choice (Relaxation Training, Behavioral Activation, or Cognitive Therapy).
- Relaxation Training only (Experimental): A 4-session telehealth Relaxation Training intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis and the cognitive behavioral model of multiple sclerosis fatigue, b) treatment rationale, c) didactic and experiential training in relaxation techniques such as diaphragmatic breathing, progressive muscle relaxation, and autogenic relaxation, and d) goal setting and problem-solving barriers to integrate relaxation practices into daily routine.
  Interventions: Behavioral: 4-session Relaxation Training
- Behavioral Activation only (Experimental): A 4-session telehealth Behavioral Activation intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, and self-monitoring activity and energy, b) treatment rationale, c) identification of values/priorities to guide activities, d) activity planning, e) goal setting and problem-solving barriers to engaging in activities.
  Interventions: Behavioral: 4-session Behavioral Activation
- Cognitive Therapy only (Experimental): A 4-session telehealth Cognitive Therapy intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, self-monitoring thoughts, and core beliefs, b) treatment rationale, c) labeling thoughts as helpful, unhelpful, or neutral, d) using distraction to cope with unhelpful thoughts, e) challenging and changing unhelpful thoughts, f) problem-solving barriers to coping with or changing unhelpful thoughts.
  Interventions: Behavioral: 4-session Cognitive Therapy
- Relaxation Training and Behavioral Activation (Experimental): 4 sessions of telehealth Relaxation Training and 4 sessions of telehealth Behavioral Activation for multiple sclerosis fatigue that are derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. Each intervention involves 4, 30-60-minute sessions delivered via phone or videoconference.
  Interventions: Behavioral: 4-session Relaxation Training; Behavioral: 4-session Behavioral Activation
- Relaxation Training and Cognitive Therapy (Experimental): 4 sessions of telehealth Relaxation Training and 4 sessions of telehealth Cognitive Therapy for multiple sclerosis fatigue that are derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. Each intervention involves 4, 30-60-minute sessions delivered via phone or videoconference.
  Interventions: Behavioral: 4-session Relaxation Training; Behavioral: 4-session Cognitive Therapy
- Behavioral Activation and Cognitive Therapy (Experimental): 4 sessions of telehealth Behavioral Activation and 4 sessions of telehealth Cognitive Therapy for multiple sclerosis fatigue that are derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. Each intervention involves 4, 30-60-minute sessions delivered via phone or videoconference.
  Interventions: Behavioral: 4-session Behavioral Activation; Behavioral: 4-session Cognitive Therapy
- Relaxation Training, Behavioral Activation, and Cognitive Therapy (Experimental): 4 sessions of telehealth Relaxation Training, 4 sessions of telehealth Behavioral Activation, and 4 sessions of telehealth Cognitive Therapy for multiple sclerosis fatigue that are derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. Each intervention involves 4, 30-60-minute sessions delivered via phone or videoconference.
  Interventions: Behavioral: 4-session Relaxation Training; Behavioral: 4-session Behavioral Activation; Behavioral: 4-session Cognitive Therapy

INTERVENTIONS:
Behavioral: 4-session Relaxation Training — A 4-session telehealth Relaxation Training intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis and the cognitive behavioral model of multiple sclerosis fatigue, b) treatment rationale, c) didactic and experiential training in relaxation techniques such as diaphragmatic breathing, progressive muscle relaxation, and autogenic relaxation, and d) goal setting and problem-solving barriers to integrate relaxation practices into daily routine.
  Arms: Relaxation Training and Behavioral Activation; Relaxation Training and Cognitive Therapy; Relaxation Training only; Relaxation Training, Behavioral Activation, and Cognitive Therapy
Behavioral: 4-session Behavioral Activation — A 4-session telehealth Behavioral Activation intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, and self-monitoring activity and energy, b) treatment rationale, c) identification of values/priorities to guide activities, d) activity planning, e) goal setting and problem-solving barriers to engaging in activities.
  Arms: Behavioral Activation and Cognitive Therapy; Behavioral Activation only; Relaxation Training and Behavioral Activation; Relaxation Training, Behavioral Activation, and Cognitive Therapy
Behavioral: 4-session Cognitive Therapy — A 4-session telehealth Cognitive Therapy intervention for multiple sclerosis fatigue that is derived from evidence-based multicomponent CBT for multiple sclerosis fatigue. The intervention is based on the cognitive behavioral model of fatigue in multiple sclerosis. The intervention involves 4, 30-60-minute sessions including the following content a) education about fatigue in multiple sclerosis, the cognitive behavioral model of multiple sclerosis fatigue, self-monitoring thoughts, and core beliefs, b) treatment rationale, c) labeling thoughts as helpful, unhelpful, or neutral, d) using distraction to cope with unhelpful thoughts, e) challenging and changing unhelpful thoughts, f) problem-solving barriers to coping with or changing unhelpful thoughts.
  Arms: Behavioral Activation and Cognitive Therapy; Cognitive Therapy only; Relaxation Training and Cognitive Therapy; Relaxation Training, Behavioral Activation, and Cognitive Therapy

SUMMARY:
This randomized controlled factorial trial will examine whether and how relaxation training, behavioral activation, and cognitive therapy improve fatigue and functioning in fatigued adults living with multiple sclerosis.

DETAILED DESCRIPTION:
Fatigue affects 80% of people with multiple sclerosis (PwMS), and nearly half report fatigue as their most disabling symptom. The cognitive behavioral model of MS fatigue theorizes that MS disease factors trigger fatigue, but fatigue is maintained or worsened by factors like daily stress and how PwMS react cognitively, behaviorally, physiologically, and emotionally to fatigue. In-person and telehealth cognitive behavioral therapy (CBT) for fatigue targets these factors and reactions and is one of the most effective treatments for MS fatigue. However, CBT is resource intensive, as it consists of multiple components (i.e., relaxation training, behavioral activation, cognitive therapy), requiring 8-16 hour-long sessions delivered by a specialized clinician. CBT has yet to be assessed via an integrated translational model that considers all stages, from intervention development to implementation. Thus, the active components of CBT for MS fatigue and their mechanisms are unclear and, despite the significant burden of MS fatigue, CBT for fatigue is not widely accessible due to various implementation barriers.

This optimization randomized controlled trial is the second aim of a research project using the Multiphase Optimization Strategy to optimize CBT for MS fatigue (1K23HD111628, Knowles, PI). This trial employs a balanced factorial design to test the main and interactive effects of the three telehealth CBT components: Relaxation Training, Behavioral Activation, and Cognitive Therapy. In this trial, each CBT component corresponds to an experimental factor that is being manipulated to obtain information about the CBT component. Each factor has two levels (Included or Excluded). The investigators are testing three factors/CBT components, yielding a 2^3 factorial trial with eight experimental conditions. Each condition corresponds to a combination of levels of the 3 factors/CBT components (e.g., a participant may be randomly assigned to a condition including zero, one, two, or three CBT components). Participants will be offered the choice of completing treatment by telephone or videoconference. Participants will complete patient reported outcome measures at pre-intervention, post-intervention, and 3 months post-intervention (follow-up). A random sample of two participants from each trial condition with at least one component will also complete qualitative interviews at post-intervention.

The overall project aims to optimize CBT for fatigue to maximize efficacy and efficiency. The project uses the Multiphase Optimization Strategy to advance scientific evidence on CBT's active components and facilitate implementation, thereby improving accessibility.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed MS diagnosis of any subtype
2. Score of 4 or higher on the Fatigue Severity Scale
3. Able to fluently converse and read in English
4. 18 years of age or older
5. Able to comply with study procedures and complete self-report measures
6. Willing to have intervention sessions audiotaped for fidelity coding
7. Has experienced fatigue for 3 or more months

Exclusion Criteria:

1. MS relapse within last 30 days (although participants will be considered eligible after the 30-day window)
2. Change in disease modifying medications (DMTs) in the prior three months (although participants will be considered eligible after the 3-month window)
3. Current suicidal ideation with intent or plan as indicated by a score of ≥1 on the Patient Health Questionnaire-9 suicide item and further assessment via the Columbia Suicide Severity Rating Scale (although individuals with suicidal ideation but no intent or plan will be considered eligible)
4. Currently engaged in psychotherapy for fatigue
5. Currently participating in another research study that could impact fatigue such as intervention studies targeting mood, energy management, exercise/physical activity, and diet (although participants can be screened for eligibility again once they have completed the other research study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 21-item self-report questionnaire assessing fatigue-related symptoms in the previous four weeks via 5-point Likert-type scale. A higher score indicates greater fatigue.
PROMIS Short Form - Ability to Participate in Social Roles and Activities | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This 8-item short form is a self-report questionnaire that assesses the perceived ability to perform one's usual social roles and activities via 5-point Likert-type scale. A lower score indicates lower ability to participate in social roles and activities.

SECONDARY OUTCOMES:
Perceived Stress Questionnaire - Tension scale | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 5-item self-report scale assessing tense disquietude, exhaustion, and the lack of relaxation via a 4-point Likert-type scale. A higher score indicates greater tension.
Behavioral Activation for Depression Scale Short Form | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 9-item self-report measure. It assess the extent to which the respondent thinks they have engaged in pleasant and/or goal-directed activity over the past week via a 7-point Likert-type scale. A higher score indicates greater behavioral activation.
Fatigue Catastrophizing Scale | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 13-item self-report questionnaire assessing negative beliefs or expectations connected to one's perceptions of fatigue via a 5-point Likert-type scale. A higher score indicates greater fatigue catastrophizing.
The Multiple Sclerosis-Fatigue Self Efficacy Scale | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 8-item self-report measure. It assesses the extent to which the respondent believes that they can manage and/or control their fatigue via a 10-point Likert-type scale. A higher score indicates greater fatigue self-efficacy.
Perceived Stress Scale | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 10-item self-report measure. It assess the extent to which the respondent perceives their life as unpredictable, uncontrollable, and overloaded via a 5-point Likert-type scale. A higher score indicates greater perceived stress.
Positive and Negative Affect Schedule | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 20-item self-report scale assessing the extent to which the respondent experiences positive and negative emotional states via a 5-point Likert-type scale. Higher Positive Affect scores indicate more positive affect, while higher Negative Affect scores indicate more negative affect.
PROMIS Emotional Distress-Depression - Short Form 4a | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This 4-item short form is a self-report questionnaire that assesses depression symptoms via 5-point Likert-type scale. A higher score indicates greater depression.
EQ-5D-5L | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 6-item measure assessing perceptions of health-related quality of life in adults. It consists of a "descriptive system" and a visual analog scale (VAS). For the descriptive system, the respondent rates five dimensions of their health state on that day - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression - by selecting the most appropriate statement that conveys their level of problem severity in each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems). Additionally, using the VAS, the respondent rates their overall health on a scale of 0 (worst imaginable health) to 100 (best imaginable health).
Global Impression of Change Scale | Collected via online survey at post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition).
  This is a single-item self-report scale that assesses the perceived intervention-related change in their activity limitations, symptoms, emotions, and overall quality of life via 7-point Likert-type scale. It has been validated in adults with multiple sclerosis.
Global Assessment of Treatment Satisfaction | Collected via online survey at post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition).
  This is a single-item self-report scale that assesses the perceived overall satisfaction with the treatment via 6-point Likert-type scale.
Treatment Recommendation Question | Collected via online survey at post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition).
  This is a single-item self-report that assesses whether a participant would recommend the intervention to a friend with MS fatigue with response options: Yes, No, Unsure, Prefer not to answer.
PROMIS Emotional Distress- Anxiety Short Form 4a | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 4-item self-report questionnaire assessing symptoms of anxiety via a 5-point Likert-type scale.
PROMIS Pain Interference Short Form 4a | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 4-item self-report questionnaire assessing pain interference via a 5-point Likert-type scale.
PROMIS Sleep Disturbance Short Form 4a | Collected via online survey at baseline/pre-treatment, post-treatment (3 days after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 4-item self-report questionnaire assessing sleep disturbance via a 5-point Likert-type scale.
Ecological Momentary Assessment of Fatigue Severity and Interference | Collected via online survey at baseline/pre-treatment, post-treatment (1 day after last treatment session or 2 months post-randomization for participants in the No Treatment condition), and 3-month follow-up.
  This is a 6-8-item measure sent 2x/day (morning and evening) for 7 days. It assesses mental and physical fatigue severity and interference on an 11-point numeric rating scale. The morning survey also assesses sleep duration as well as sleep quality via 2 questions rated on a Likert-type scale. The evening survey also assess perceived fatigue management efforts via 2 questions rated on a Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Knowles, PhD, Principal Investigator — University of Washington
Locations (1):
- Multiple Sclerosis Center at UW Medical Center - Northwest, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make available to interested researchers a data file containing de-identified data used for each published article at the time the article is accepted for publication. The data will be de-identified to remove any variables from which it would be possible to identify any individual participants. Specifically, the investigators will create a data file that includes all variables used in the published article and a list of the variables in the data file (along with variable labels) and send to investigators who request the data a copy of: (1) the published article (which will describe the source of the data); (2) the variable list/variable labels; and (3) the dataset (as an SPSS.sav file). Note, though, even though any data files that the investigators share will be stripped of identifiers prior to release for sharing, it remains possible those who access the data could potentially use deduction to identify participants with unusual characteristics or combinations o
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data used for the analyses for any papers published will become available to interested researchers by request after that article is published. Those data will continue to be available for at least five years following the publication of the article.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- See also: Study Website — https://uwmsrehabwell.org/cbt-for-ms-fatigue-2/